CLINICAL TRIAL: NCT06646783
Title: Clinical Study of 68GA-labeled Claudin 18.2 Developer Combined with PET/CT for Imaging of Gastric or Gastroesophageal Junction Adenocarcinoma and Pancreatic Cancer
Brief Title: Phase IIT Trial of SNA014
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: SmartNuclide Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: [68Ga]Ga-NODAGA-SNA014
Record Dates: First submitted 2024-10-10; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Adenocarcinoma of the Stomach; Adenocarcinoma of GE Junction; Pancreatic Cancer Stage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- dose escalation (Experimental): subgroups mass does escalation
  Interventions: Drug: [68Ga]Ga-NODAGA-SNA014

INTERVENTIONS:
Drug: [68Ga]Ga-NODAGA-SNA014 — Perform whole-body PET/CT scans on the subjects at 30 minutes (± 5 minutes), 60 minutes (± 10 minutes), 120 minutes (± 20 minutes), and 240 minutes (± 30 minutes) after administration. Among them, PET scanning can be performed on 1-2 subjects in a certain dose group or each dose group for 30-60 minutes. Among the four CT scans, one CT scan is a conventional low-dose CT scan (120mA), and the remaining three are extremely low-dose CT scans (10-20mA). The main researchers and nuclear medicine physicians can decide whether to change the subsequent image acquisition time and duration of the subjects based on the image information obtained from the enrolled subjects.

SUMMARY:
68Ga labeled Claudin 18.2 contrast agent combined with PET/CT for gastric or gastroesophageal junction

ELIGIBILITY:
Inclusion Criteria:

* Age range of 18 to 75 years old (including boundary values);
* Individuals with behavioral capacity who voluntarily participate in this clinical study and sign an informed consent form (ICF);
* Diagnosed G/GEJ adenocarcinoma and pancreatic cancer;
* Gastroscopy/CT/MRI/PET-CT examination results within the past month (if any);
* Pathological test results and Claudin18.2 immunohistochemistry results within the past year (if available).

Exclusion Criteria:

* Merge patients with other clearly diagnosed malignant tumors:
* Uncontrolled severe infections or individuals with other serious illnesses;
* Those with an expected survival period of less than or equal to three months;
* Pregnant or lactating patients, as well as reproductive age patients who refuse to take appropriate contraceptive measures during this trial;
* investigators determine that patients who are not suitable to participate in this study;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-10-20 (Estimated); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
Biological distribution characteristics | 1week
  Evaluate the biological distribution characteristics of important organs in the subjects.
  * Draw the Volume of Interest (VOI) of the subject's vital organs and calculate the Percentage of Injected Activity (IA) of the vital organs
  * Using PMOD software, manually draw regions of interest (VOI) on PET/CT images of the liver, spleen, normal stomach, heart, bone marrow, kidneys, and other areas to obtain the cumulative radioactive activity of these regions. Divide the cumulative radioactive activity by the injection dose to obtain the percentage of injection activity (% IA).
Safety tolerance characteristics | hrough study completion, an average of 1 year
  AE/SAE/SUSAR

SECONDARY OUTCOMES:
Metabolic Dynamics Evaluation and Radiation Dose | 1 day
  Detect the radiation dose of whole blood and serum of the subjects, and calculate the absorbed dose of important organs

OTHER OUTCOMES:
Exploring the targeting ability of CLDN18.2 | 1month
  Correlation analysis between PET/CT imaging features of target lesions (SUVmax, SUV mean, target to body ratio, etc.) and CLDN18.2IHC expression level (if any)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Jiangsu, Province, China

IPD SHARING:
Plan to Share IPD: Yes